CLINICAL TRIAL: NCT00230945
Title: Psychobiological Pathways: Osteoarthritis Interventions
Brief Title: Couples-Oriented Psychosocial Intervention for Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Lynn M. Martire, Ph.D., Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50 HL65111-65112--2; P50HL065111 (NIH)
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patient-oriented education and support intervention
  Interventions: Behavioral: education and support intervention
- 2 (Experimental): Couple-oriented education and support intervention
  Interventions: Behavioral: education and support intervention

INTERVENTIONS:
Behavioral: education and support intervention — The patient-oriented education and support intervention (PES) is based on the Arthritis Self-Management Program, a group intervention that consists of 6 weekly 2 hour sessions shown to successfully reduce pain severity and depressive symptomatology and to enhance a sense of efficacy in managing arthritis pain and other symptoms. The couple-oriented education and support intervention (CES) is a group education and support intervention that consisted of 6 weekly 2 hour sessions attended by individuals with OA and their spouses. All components of the PES are covered in the CES using the standard format, and topics are framed as couples' issues whenever possible.

SUMMARY:
The purpose of this study is to determine if osteoarthritis patients and their spouses experience greater health benefits from a couples-oriented psychosocial intervention than a patient-oriented psychosocial intervention, and to determine if each intervention is more beneficial than patient usual medical care.

DETAILED DESCRIPTION:
The patient-oriented education and support intervention (PES) is based on the Arthritis Self-Management Program, a group intervention that consists of 6 weekly 2 hour sessions shown to successfully reduce pain severity and depressive symptomatology and to enhance a sense of efficacy in managing arthritis pain and other symptoms. The PES specifically focuses on self-management of arthritis and no spouses, family members, or friends participate in PES sessions. Major components of the sessions include information regarding the etiology and treatment of arthritis, self-management strategies for managing pain and strengthening joints, the benefits of exercise, communication skills, and ways to effectively cope with negative emotions. At the end of each weekly session, each participant sets a health-related goal (e.g., walk for exercise three times over the next week). At the beginning of the next session each participant reports on his or her success in meeting this goal and receives feedback from the group. Participants in the PES are encouraged to communicate with, and be a source of support to, one another both within and outside the sessions. The PES facilitator is an individual who was trained by staff of the Arthritis Foundation to lead the Arthritis Self-Management Program and who follows a detailed intervention manual created for this Program and for the present study.

The couple-oriented education and support intervention (CES) is a group education and support intervention that consisted of 6 weekly 2 hour sessions attended by individuals with OA and their spouses. All components of the PES are covered in the CES using the standard format, and topics are framed as couples' issues whenever possible. An overarching framework introduced in the first session of the CES is that pain is a complex experience which can be influenced by thoughts, feelings, and behaviors; spouses can influence and be affected by these same thoughts, feelings, and behaviors; and spouses' concerns and experiences as support providers are important to address. Each of the next 5 sessions is supplemented by a component that was linked to a topic covered in the PES and explicitly extended to couples. For example, a topic of the third session of the PES deals with managing fatigue and the supplemental component for this session provides information on the most effective and ineffective strategies for requesting spousal assistance (e.g., verbal versus nonverbal pain expression and the need to be clear about help needed) and providing spousal assistance (e.g., consider timing and amount of assistance desired). The supplemental components for the 4 remaining sessions address spouse encouragement and practice of cognitive or behavioral pain management strategies (e.g., distraction and progressive muscle relaxation); supportive and unsupportive spousal communications; reducing negative emotional contagion between partners; and couples' strategies for managing medications. At the end of each weekly session of the CES, each individual with OA and his or her spouse sets health-related goals for the following week and their success in meeting these goals iss reviewed with the group at the beginning of the next session. Spouses are instructed to set goals that were facilitative of their partners' goals whenever possible. Couples in the CES are encouraged to communicate with, and be a source of support to, one another both within and outside the course. The CES facilitator is trained in the Arthritis Self-Management Program by staff of the Arthritis Foundation and in the couples materials by study investigators, and follows a detailed intervention manual.

The no-treatment control group received usual medical care only.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis in back, hips, and/or knees(patients) married and co-residing age 50 or older pain of at least moderate intensity difficulty with at least one instrumental ADL receiving help from spouse w/ at least one instrumental IADL

Exclusion Criteria:

* fibromyalgia or rheumatoid arthritis taken Arthritis Self-Help Course in past 5 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2000-01; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
patient pain, disability, and depressive symptoms. spouse stress and negative affect | 6 months

SECONDARY OUTCOMES:
positive affect, exercise, spousal support and critical attitudes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M. Martire, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States